CLINICAL TRIAL: NCT06252532
Title: Modulating Oscillations and Working Memory in Patients With Subdural Electrodes
Brief Title: Causal Role of Top-Down Theta Oscillations in Prioritization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-1652; 5R01MH124387 (NIH)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Working Memory; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Frontal Stimulation (Active Comparator): Direct Cortical Stimulation (DCS) in alpha and theta frequencies is applied through electrodes located in the frontal cortex.
  Interventions: Device: Direct cortical stimulation (DCS) Alpha; Device: Direct cortical stimulation (DCS) Theta; Device: Sham Direct cortical stimulation (DCS)
- Frontal Parietal Stimulation (Sham Comparator): Direct Cortical Stimulation (DCS) in in-phase and anti-phase theta frequencies is applied through electrodes located in the frontal and parietal cortex.
  Interventions: Device: Sham Direct cortical stimulation (DCS); Device: Direct cortical stimulation (DCS) In-Phase Theta; Device: Direct cortical stimulation (DCS) Anti-Phase Theta

INTERVENTIONS:
Device: Direct cortical stimulation (DCS) Alpha — Rhythmic alpha stimulation
  Other Names: CereStim M96
  Arms: Frontal Stimulation
Device: Direct cortical stimulation (DCS) Theta — Rhythmic theta stimulation applied
  Other Names: CereStim M96
  Arms: Frontal Stimulation
Device: Sham Direct cortical stimulation (DCS) — Arrhythmic stimulation paradigm applied
  Other Names: CereStim M96
Device: Direct cortical stimulation (DCS) In-Phase Theta — Rhythmic in-phase theta stimulation applied
  Other Names: CereStim M96
  Arms: Frontal Parietal Stimulation
Device: Direct cortical stimulation (DCS) Anti-Phase Theta — Rhythmic anti-phase theta stimulation applied
  Other Names: CereStim M96
  Arms: Frontal Parietal Stimulation

SUMMARY:
Purpose: The purpose of this pilot study is to investigate the dynamics between theta and alpha oscillations in the control of working memory. These findings will be informative of what types of brain stimulation are most effective at modulating brain activity. Deep brain stimulation and transcranial magnetic stimulation are used for an increasing number of neurological and psychiatric disorders. Participants: Eligible participants are patients who have previously had electrodes implanted to monitor epilepsy (outside of research activity). 50 participants will be recruited, 25 participants for each phase of the study. Procedures (methods): The participants will perform a cognitive control task. During the task, rhythmic trains of direct cortical stimulation will be delivered to the frontal cortex alone or to the frontal and parietal cortex. Electrocorticography will be collected concurrent with stimulation.

DETAILED DESCRIPTION:
The aim of this study is to investigate the causal role of functional interactions between frontal-theta dependent selection processes and posterior-alpha dependent suppression processes in the context of cognitive control by targeting theta and alpha oscillations in frontal and parietal cortex separately in phase one of the experiment. Theta and alpha oscillations are hypothesized to play complementary roles such that theta oscillations are excitatory (related to active processing) whereas alpha oscillations are inhibitory (related to suppression of processing).

Thus, the investigators hypothesize that rhythmic brain stimulation can be used to drive activity in opposite directions. In the second phase of the experiment the investigators target functional connectivity between these regions. In particular, theta oscillations are hypothesized to play a critical role in orchestrating the prioritization and suppression of information across the cerebral cortex. Thus, the investigators hypothesize that in-phase theta frequency connectivity will be causally related to working memory success, but alpha frequency connectivity will be inconsequential and anti-phase theta connectivity will be detrimental. Together these findings suggest an overall model by which the amplitude of theta oscillations in prefrontal and the amplitude of alpha oscillations in parietal play a causal role in prioritization and suppression respectively, but functional connectivity between frontal and parietal cortex within the theta frequency band alone is critical to these cognitive processes. This experiment is of critical importance to the design of future interventions that use brain stimulation for the treatment of psychiatric and neurological disorders. For example, the use of frequency specific brain stimulation is key to controlling the impact of brain stimulation on neural activity. Design considerations like this one might be fundamental to improving the efficacy of future interventions such as the use of deep brain stimulation for the treatment of Parkinson's disease and for the use of transcranial magnetic stimulation for the treatment of major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* History of medically intractable epilepsy
* Speak and understand English
* For the stimulation session, the participant must have electrodes in the relevant locations

Exclusion Criteria:

* Current diagnosis of other neurological illnesses including ischemic stroke, intracerebral hemorrhage, brain neoplasm
* Major systemic illness
* Severe cognitive impairment - diagnosed by clinician in neuropsychiatric evaluation
* Severe psychiatric illness
* Excessive use of alcohol or other substances
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Working Memory Task Performance - Pashler's working memory capacity metric (k) | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  The participant will be presented with three colored squares in both visual fields during a practice session. Then the participant is presented with an informative retro-cue, an arrow to the left or right, that is 100% predictive of the upcoming probe, or an uninformative neural cue, an arrow pointing in both directions. Finally, in the probe epoch participants are presented with an array of squares on the left or the right side of the screen. Participants must determine if the array of colored squares is the same or different from those held in memory. Performance will be defined as: k=N*(HR*FA)/(1-FA) where N is the number of the items that are held in memory. HR is the hit rate defined as the percent correct for trials where the probe does not match the encoding array. FA is the false alarm rate defined as the percent incorrect for trials where the probe does match the encoding array.
Change in Working Memory Task Performance - Reaction Time | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  The participant will be presented with three colored squares in both visual fields during a practice session. Then the participant is presented with an informative retro-cue, an arrow to the left or right, that is 100% predictive of the upcoming probe, or an uninformative neural cue, an arrow pointing in both directions. Finally, in the probe epoch participants are presented with an array of squares on the left or the right side of the screen. Participants must determine if the array of colored squares is the same or different from those held in memory. Reaction times will be quantified in milliseconds.
Intracranial EEG Multi-taper fft | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  Time-frequency analysis of electrophysiology data will be performed using methods like multi-taper fft. This will be compared between sham (arrhythmic) and stimulation trials to identify if stimulation enhances neuronal entrainment.
Intracranial EEG weighted phase lag index (wPLI) | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  Functional connectivity will be measured using weighted phase lag index (WPLI). To calculate WPLI, first Morlet wavelet convolution is performed to extract instantaneous phase and amplitude for the frequency of interest for the two target sites. Next, the cross-spectral density is calculated (one signal multiplied by the complex conjugate of the other). From the cross-spectral density the imaginary component of the resulting signal is extracted. Then those imaginary values are averaged over the time frame of instance (here, the second half of the stimulation train). Finally, the magnitude of the resulting vector is taken to be the wPLI. This metric quantifies the consistency of phase lag between the two target regions and is weighted towards signals with a 90 or 270 degree offset to address a common confound in electrophysiology, volume conduction.

SECONDARY OUTCOMES:
Intracranial EEG Wavelets | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  Spectral analysis and functional connectivity analysis of electrophysiology data will be performed using methods like wavelets. This will be compared between sham (arrhythmic) and stimulation trials to identify if stimulation enhances neuronal entrainment.
Intracranial EEG phase locking | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  Spectral analysis and functional connectivity analysis of electrophysiology data will be performed using methods like phase locking. This will be compared between sham (arrhythmic) and stimulation trials to identify if stimulation enhances neuronal entrainment.
Intracranial EEG Granger causality | During the 1- to 1.5-hour test at Baseline and Stimulation Session conducted over a 1 to 2 day period
  Spectral analysis and functional connectivity analysis of electrophysiology data will be performed using methods like Granger causality. This will be compared between sham (arrhythmic) and stimulation trials to identify if stimulation enhances neuronal entrainment.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Alagapan S, Riddle J, Huang WA, Hadar E, Shin HW, Frohlich F. Network-Targeted, Multi-site Direct Cortical Stimulation Enhances Working Memory by Modulating Phase Lag of Low-Frequency Oscillations. Cell Rep. 2019 Nov 26;29(9):2590-2598.e4. doi: 10.1016/j.celrep.2019.10.072. PMID 31775030
- [Background] Alagapan S, Lustenberger C, Hadar E, Shin HW, Frӧhlich F. Low-frequency direct cortical stimulation of left superior frontal gyrus enhances working memory performance. Neuroimage. 2019 Jan 1;184:697-706. doi: 10.1016/j.neuroimage.2018.09.064. Epub 2018 Sep 27. PMID 30268847